CLINICAL TRIAL: NCT04542889
Title: Study of the Coronary Microcirculation After Primary Angioplasty : Analysis of Absolute Coronary Blood Flow Rates and Resistance, Index of Microcirculatory Resistance and Comparison With Magnetic Resonance Imaging
Brief Title: Coronary Microcirculation Assessment After Primary Angioplasty in Myocardial Infarction
Acronym: NATHANAEL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of principal investigator
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190831; 2019-A02413-54 (Other: IDRCB)
Record Dates: First submitted 2020-03-06; First posted 2020-09-09 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: Coronary physiology; Coronary microvascular circulation; STEMI; Microvascular Obstruction; No Reflow; Rayflow®; Absolute coronary resistance; IMR
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Absolute coronary resistances and IMR after angioplasty (Experimental): Patients with STEMI by acute occlusion of a large caliber coronary artery that had been admitted to hospital less than 12 hours and revascularized by primary angioplasty with good final result.
  Interventions: Diagnostic Test: Absolute coronary flow and resistance measurements; Diagnostic Test: IMR measurement

INTERVENTIONS:
Diagnostic Test: Absolute coronary flow and resistance measurements — Thermodilution-based measurements of absolute coronary resistances using the FFR pressure guide (PressureWire® Certus® from St Jude Medical Abbott) and the Rayflow® microcatheter (Hexacath, Paris, France).
Diagnostic Test: IMR measurement — IMR measurement by thermodilution using the St Jude pressure guide.

SUMMARY:
In the management of acute myocardial infarction treated with primary angioplasty, despite effective epicardial clearance obtained in 95% of cases, microvascular obstruction (MVO) in the damaged territory concerns 50% of patients. The Index of Microvascular Resistance (IMR) allows early assessment of the microcirculatory state during the angioplasty procedure. A value of IMR>40 indicates MVO and is correlated with morbi-mortality. A new method for immediate evaluation of MVO using thermodilution with a new Rayflow® microcatheter has been described: it no longer allows the estimation but the measurements of absolute coronary resistance and coronary flow. We hypothesize that these measurements allows a better evaluation of the microcirculatory state after primary angioplasty, comparing to IMR.

The main objective is to study the diagnostic performance of Rayflow® to predict MVO - no reflow (NR) - in ST-Elevation Myocardial Infarction (STEMI) patients in order to determine an absolute coronary resistance threshold by thermodilution for early diagnosis of MVO.

The main secondary objectives will be to compare the different microcirculatory assessment parameters with each other, not indexed and indexed to the myocardial mass at risk (coronary resistance, IMR, CFR, Resistance Reserve Ratio) and to establish a link between high resistance or IMR and the occurrence of rhythm disorders at D1, D2 and D3.

DETAILED DESCRIPTION:
All patients presenting for STEMI by occlusion of a proximal coronary artery, vascularizing a large volume of myocardium corresponding to an APPROACH score> 21, in the first 12 hours following the onset of chest pain, will be included.

Data relating to medical history, lifestyle (sedentary lifestyle, smoking, drug use), cardiovascular risk factors will be collected.

The management of acute coronary syndrome will be carried out in accordance with the European Society of Cardiology guidelines of 2015. An emergency coronary angiography will be used to revascularise the patient as indicated. Thromboaspiration, stenting, antithrombotic agents and other treatments will be administered according to angiographic and clinical criteria.

The FFR guide (PressureWire® Certus® from St Jude Medical Abbott) will be used to make pressure and temperature measurements. It has been used in daily practice since the FAME study in 2011 to guide the therapeutic decision in patients with an intermediate lesion.

An injected cardiac magnetic resonance imaging (MRI) will be performed between 48 hours and 7 days following the infarction in accordance with current practices.The initial trans-thoracic ultrasonography as well as the various blood samplings will be performed according to standard practice.

The Rayflow® microcatheter will be used to allow the optimal delivery of physiological saline solution into the studied artery. It will be mounted on the FFR guide already in place as part of the angioplasty procedure. Bayer's Medrad® Mark 7 Arterion® infuser will be used to deliver saline continuously at a flow rate of 15-20 mL/min through the Rayflow® microcatheter

ELIGIBILITY:
Inclusion Criteria:

* Acute ST + coronary syndrome seen within 12 hours after the initial pain: ST offset in 2 contiguous leads ≥ 1mm or ≥ 2mm in precordial or inaugural left branch block, permanent or transient with chest pain > 20 min
* Patient with an indication for emergency coronary angiography with angioplasty
* Acute occlusion of a large caliber artery corresponding to an APPROACH score ≥21: proximal or mean anterior interventricular artery, proximal circumflex artery or proximal right coronary artery
* Final Thrombolysis In Myocardial Infarction (TIMI) of 2 or 3 at the end of the angioplasty procedure regardless of the initial TIMI score
* Free and informed written consent to participate in the study

Exclusion Criteria:

* Known history of infarction in the same territory : STEMI or NSTEMI (angioplasty programmed for angina does not constitute a criterion for non-inclusion)
* Haemodynamic instability requiring the initial use of vasopressive amines or circulatory assistance (counterpulse balloon or extracorporeal membrane oxygenation) or mechanical ventilation (a recovered cardiopulmonary arrest does not constitute an exclusion criterion)
* Technical impossibility of performing IMR or Rayflow® measurements (tortuous or calcified artery)
* Persistent high-grade atrioventricular block after primary angioplasty
* Cardiomyopathy or severe valvulopathy which can induce microcirculatory abnormalities (congenital heart diseases, dilated cardiomyopathy, cardiac amyloidosis, hypertrophic heart disease, mitral regurgitation, aortic regurgitation, tricuspid regurgitation or pulmonary regurgitation grade 3 or 4, tight aortic stenosis or pulmonary stenosis with average gradient > 40 mmHg or vmax > 4m/sec , tight mitral stenosis or tricuspid stenosis with average gradient > 10mmHg)
* Contraindication to performing cardiac MRI: wearing a pacemaker, intracerebral clip, intraocular foreign body, neurostimulator, severe renal failure with glomerular filtration rate < 30 mL/min, body weight > 150 kg
* Age < 18 years
* Pregnant or breastfeeding woman
* Inclusion in another research protocol < 30 days
* Patient not affiliated to a social security scheme
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Absolute coronary resistance | Immediately after angioplasty
  Threshold value correlated with microvascular obstruction on magnetic resonance imaging (MRI)
Microvascular obstruction on MRI | Day 7
  Establishment of a correlation between absolute coronary resistance and microvascular obstruction on MRI

SECONDARY OUTCOMES:
Index of microvascular resistance | Immediately after angioplasty
  Threshold value correlated with microvascular obstruction on MRI
Mean value of absolute coronary resistances corresponding to an IMR > 40 | Immediately after angioplasty
  Establishment of a relationship between absolute coronary resistances and IMR
Microvascular obstruction in patients with IMR > 40 | Day 7
  Establishment of a correlation between an IMR> 40 and the presence and the degree of microvascular obstruction as meaasured by cardiac MRI of the of infarcted area
Absolute coronary resistance indexed to the myocardial mass | Immediately after angioplasty
  Establishment of a correlation between the indexed absolute coronary resistance and the presence and the degree of microvascular obstruction on cardiac MRI
IMR indexed to the myocardial mass | Immediately after angioplasty
  Establishment of a correlation between the indexed IMR and the presence and the degree of microvascular obstruction on cardiac MRI
Occurrence of early ventricular rhythm disorders | Day 3
  Establishment of a correlation between the absolute coronary resistances and IMR and the early ventricular rhythm disorders

CONTACTS AND LOCATIONS:
Overall Officials: Georgios SIDERIS, MD, Principal Investigator — APHP, Lariboisière Hospital, Cardiology Department
Locations (1):
- APHP, Lariboisière Hospital, Cardiology Department, Paris, France